CLINICAL TRIAL: NCT04169191
Title: Treatment of Neonatal Encephalopathy With Oral Sildenafil Suspension to Repair Brain Injury Secondary to Birth Asphyxia: An Open-label Dose-finding Clinical Trial (Phase Ib Study)
Brief Title: Sildenafil to Repair Brain Injury Secondary to Birth Asphyxia
Acronym: SANE-02
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Pia Wintermark, Associate Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SANE-02
Record Dates: First submitted 2019-10-01; First posted 2019-11-19 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Birth Asphyxia
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: 3+3 design to escalate the sildenafil dose up to 6 mg/kg/day (3mg/kg/dose q12h)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sildenafil (Experimental)
  Interventions: Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil Citrate — Cohort 1 of 3-6 neonates: 1st dose of 2mg/kg/dose, 2nd dose of 2.5 mg/kg/dose, and subsequent doses of 2.5mg/kg/dose q12h (= 5 mg/kg/day from dose #2) Cohort 2 of 3-6 neonates: 1st dose of 2mg/kg/dose, 2nd dose of 2.5 mg/kg/dose, 3rd dose of 3mg/kg/dose, and subsequent doses of 3mg/kg/dose q12h (= 6 mg/kg/day from dose #3) dose expansion phase in up to 5-15 asphyxiated neonates

SUMMARY:
The investigators will determine the maximum tolerable dose of sildenafil and establish the pharmacokinetic and pharmacodynamic profile of sildenafil in human asphyxiated neonates treated with hypothermia. They will use a 3+3 design to escalate the sildenafil dose up to 6 mg/kg/day (3mg/kg/dose q12h) in asphyxiated neonates demonstrating brain injury despite hypothermia treatment and assess whether we observe any beneficial effects of sildenafil on their brain and cardiopulmonary hemodynamics, without causing serious adverse events

ELIGIBILITY:
Inclusion Criteria:

* Male and female neonates meeting the criteria for induced hypothermia:

  * Gestational age ≥ 36 weeks and birth weight ≥ 1800 g;
  * Evidence of fetal distress, i.e., history of an acute perinatal event, cord pH ≤ 7.0 or base deficit ≤ - 16 mEq/L;
  * Evidence of neonatal distress, such as an Apgar score ≤ 5 at 10 minutes, postnatal blood gas pH obtained within the first hour of life ≤ 7.0 or base deficit ≤ - 16 mEq/L, or a continued need for ventilation initiated at birth and continued for at least 10 minutes;
  * Evidence of moderate to severe neonatal encephalopathy by an abnormal neurological exam and/or an amplitude-integrated electroencephalogram (aEEG).
* Evidence of brain injury on a brain magnetic resonance imaging (MRI) performed on day 2 of life.

Exclusion Criteria:

* Neonates with complex congenital heart disease
* Neonates with cerebral malformations
* Neonates with genetic syndrome
* Neonates with intraventricular and/or intraparenchymal hemorrhage on MRI performed on day 2 of life

Ages: 0 Days to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Death | within first 10 days of life
  Number of participants with death
Hypotension | within first 10 days of life
  Number of participants with hypotension

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | within first 10 days of life
  Peak Plasma Concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Derived] Wintermark P, Lapointe A, Altit G, Steinhorn R, Rampakakis E, Meid AD, Burhenne J, Bajraktari-Sylejmani G, Khairy M, Adamo MT, Gilbert G, Toffoli D, Zavalkoff S, Luu TM, Hailu E, Haefeli WE. Testing Higher Doses of Sildenafil to Repair Brain Injury Secondary to Birth Asphyxia: An Open-Label Dose-Finding Phase 1b Clinical Trial-Sildenafil Administration to Treat Neonatal Encephalopathy-Study 02. J Pediatr. 2025 Oct;285:114701. doi: 10.1016/j.jpeds.2025.114701. Epub 2025 Jun 23. PMID 40562301